CLINICAL TRIAL: NCT06990867
Title: Optimizing Reperfusion to Improve Outcomes and Neurologic Function (ORION): A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group, Phase 2/3 Study to Evaluate the Efficacy and Safety of JX10 in Acute Ischemic Stroke With Late Presentations
Brief Title: Optimizing Reperfusion to Improve Outcomes and Neurologic Function
Acronym: ORION
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JX10002
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
Keywords: reperfusion; ORION; Acute Ischemic Stroke; Late Presentation; JX10; thrombolytic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 - JX10 (1mg/kg) (Experimental)
  Interventions: Drug: JX10
- Part 1 - JX10 (3mg/kg) (Experimental)
  Interventions: Drug: JX10
- Part 1 - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- JX10 Part 2 - (1 or 3 mg/kg) (Experimental)
  Interventions: Drug: JX10
- Part 2 - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JX10 — JX10 is a thrombolytic agent.
  Arms: JX10 Part 2 - (1 or 3 mg/kg); Part 1 - JX10 (1mg/kg); Part 1 - JX10 (3mg/kg)
Drug: Placebo — Placebo is being used as the comparator.
  Arms: Part 1 - Placebo; Part 2 - Placebo

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of JX10 versus placebo in participants with Acute Ischemic Stroke (AIS) who present for care within 4.5 to 24 hours.

The main question the study aims to answer are:

1. JX10 improves functional outcomes as measured by the modified Rankin Scale score when compared with placebo following AIS.
2. Risk of symptomatic intracranial hemorrhage of JX10 in participants with AIS.

During Part 1, participants will be randomized to JX 10 (1mg/kg, 3 mg/kg) or placebo. During Part 2, participants will receive JX10 (optimal dose chosen from Part 1) or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 90 years old.
2. Acute ischemic stroke with compatible clinical presentation and symptomatic high grade or complete occlusion of the intracranial internal carotid, M1, M2 or distal branches of the middle cerebral artery (MCA), anterior cerebral artery (ACA), or posterior cerebral artery (PCA).
3. Radiographic evidence of salvageable tissue.
4. Pre-treatment score of NIHSS ≥ 5.

Exclusion Criteria:

1. Radiographic findings pre-randomization of any of the following:

   1. Large core infarction, or
   2. Occlusion in more than 1 vascular territory, or
   3. Significant mass effect or clinically significant cerebral edema, or
   4. Evidence of acute intracranial or extracranial hemorrhage, intracranial tumor (except small meningioma), neoplasm, or arteriovenous malformation), or
   5. Clinical history, past imaging, or clinical judgement suggests that the intracranial occlusion is chronic.
2. Medical history or active clinically significant bleeding, lesions, or conditions (at the investigator's judgement) considered to be of significant risk for major bleeding.
3. Severe, uncontrolled hypertension (systolic blood pressure ≥ 185 mmHg or diastolic blood pressure ≥ 110 mmHg) that cannot be controlled with antihypertensive therapy.
4. Known bleeding diathesis (hereditary or acquired) or any significant coagulopathy. Specifically, platelet count < 100,000/μL, international normalized ratio > 1.7, aPTT > 40 seconds, or prothrombin time > 15 seconds.
5. Major trauma, surgery, or invasive procedures.
6. Pre-existing medical, neurological, or psychiatric disease that would confound the neurological or functional evaluations of this study.
7. Pre-treatment blood glucose > 400 mg/dL (22.20 mmol/L) or Pre-treatment blood glucose < 50 mg/dL (2.78 mmol/L) unless it is corrected prior to study treatment administration. Participants with subsequently normalized blood glucose levels may be considered for inclusion, per Investigator judgement.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Proportion of participants with no or minimal symptoms (mRS score 0-1) at 90 days | 90 days
Safety: Incidence of symptomatic intracranial hemorrhage within 36 hours post-randomization | Within 36 hours post-randomization

SECONDARY OUTCOMES:
Ordinal mRS score (0-6), based on a 6-point ordinal scale at 90 days | 90 days
Proportion of participants with functional independence at 90 days | 90 days
  Functional independence: mRS score 0-2
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 90 days
Incidence of major bleeding within 24 hours and 14 days of study treatment | Within 24 hours and 14 days of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Senior Director, Clinical Operations, Study Director — Corxel Pharmaceuticals
Locations (75):
- United States (17):
  - Corxel Investigational Site, Long Beach, California
  - Corxel Investigational Site, Sacramento, California
  - Corxel Investigational Site, Colorado Springs, Colorado
  - Corxel Investigational Site, Washington D.C., District of Columbia
  - Corxel Investigational Site, Delray Beach, Florida
  - Corxel Investigational Site, Chicago, Illinois
  - Corxel Investigational Site, Wichita, Kansas
  - Corxel Investigational Site, Baltimore, Maryland
  - Corxel Investigational Site, Kalamazoo, Michigan
  - Corxel Investigational Site, Traverse City, Michigan
  - Corxel Investigational Site, St Louis, Missouri
  - Corxel Investigational Site, Great Neck, New York
  - Corxel Investigational Site, New York, New York
  - Corxel Investigational Site, Toledo, Ohio
  - Corxel Investigational Site, Tulsa, Oklahoma
  - Corxel Investigational Site, Dallas, Texas
  - Corxel Investigational Site, Houston, Texas
- Corxel Investigational Site, Ghent, Belgium
- Bulgaria (5):
  - Corxel Investigational Site, Blagoevgrad
  - Corxel Investigational Site, Burgas
  - Corxel Investigational Site, Pleven
  - Corxel Investigational Site, Plovdiv
  - Corxel Investigational Site, Sofia
- Canada (2):
  - Corxel Investigational Site, Edmonton
  - Corxel Investigational Site, Kingston
- China (13):
  - Corxel Investigational Site, Baotou
  - Corxel Investigational Site, Beijing
  - Corxel Investigational Site, Changchun
  - Corxel Investigational Site, Guangzhou
  - Corxel Investigational Site,, Harbin
  - Corxel Investigational Site, Harbin
  - Corxel Investigational Site, Kaili
  - Corxel Investigational Site, Linfen
  - Corxel Investigational Site, Shanghai
  - Corxel Investigational Site, Shenyang
  - Corxel Investigational Site, Suzhou
  - Corxel Investigational Site, Weifang
  - Corxel Investigational Site, Xuzhou
- Germany (3):
  - Corxel Investigational Site, Altenburg
  - Corxel Investigational Site, Leipzig
  - Corxel Investigational Site, Lübeck
- Greece (3):
  - Corxel Investigational Site, Athens
  - Corxel Investigational Site, Chaïdári
  - Corxel Investigational Site, Thessaloniki
- Italy (2):
  - Corxel Investigational Site, Pavia
  - Corxel Investigational Site, Roma
- Japan (7):
  - Corxel Investigational Site, Fukuoka
  - Corxel Investigational Site, Hyōgo
  - Corxel Investigational Site, Kamakura
  - Corxel Investigational Site, Mitaka
  - Corxel Investigational Site, Miyagi
  - Corxel Investigational Site, Yamagata
  - Corxel Investigational Site, Yamaguchi
- Latvia (2):
  - Corxel Investigational Site, Daugavpils
  - Corxel Investigational Site, Riga
- Lithuania (2):
  - Corxel Investigational Site, Kaunas
  - Corxel Investigational Site, Vilnius
- Corxel Investigational Site, Kuching, Malaysia
- Portugal (2):
  - Corxel Investigational Site, Braga
  - Corxel Investigational Site, Loures
- Serbia (4):
  - Corxel Investigational Site, Belgrade
  - Corxel Investigational Site, Kragujevac
  - Corxel Investigational Site, Niš
  - Corxel Investigational Site, Novi Sad
- Corxel Investigational Site, Seoul, South Korea
- Spain (8):
  - Corxel Investigational Site, A Coruña
  - Corxel Investigational Site, Albacete
  - Corxel Investigational Site, Barcelona
  - Corxel Investigational Site, Girona
  - Corxel Investigational Site, Madrid
  - Corxel Investigational Site, Málaga
  - Corxel Investigational Site, Seville
  - Corxel Investigational Site, Valencia
- Thailand (2):
  - Corxel Investigational Site, Bangkok
  - Corxel Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: No